CLINICAL TRIAL: NCT02617784
Title: A Single Center, Open Label, Multiple-Dose Oral Oseltamivir Suspension Study in End-Stage-Renal Disease (ESRD) Patients on Hemodialysis (HD) and Continuous Ambulatory Peritoneal Dialysis (CAPD)
Brief Title: A Multiple-Dose Study of Oral Oseltamivir in Participants on Hemodialysis (HD) and Continuous Ambulatory Peritoneal Dialysis (CAPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP16472
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Oseltamivir

ARMS (2):
- Regimen A: Oseltamivir with HD (Experimental): Participants will receive 30 milligrams (mg) of oseltamivir via oral suspension approximately 1 hour after alternating HD sessions. Sessions will occur three times per week within the 6.5-week study period, and participants will receive a total of 9 doses of oseltamivir.
  Interventions: Drug: Oseltamivir
- Regimen B: Oseltamivir with CAPD (Experimental): Participants will receive 30 mg of oseltamivir via oral suspension once weekly after dialysis exchange. CAPD sessions will occur four times every 24 hours, and participants will receive a total of 6 doses of oseltamivir within the 6-week study period.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir will be given as marketed oral suspension, 30 mg after HD or CAPD treatment.
  Other Names: Tamiflu

SUMMARY:
This study is designed to assess the pharmacokinetics (PK) and safety of oseltamivir and its metabolite oseltamivir carboxylate in participants undergoing routine HD and CAPD for end-stage renal disease (ESRD). Participants will receive 6.5 and 6 weeks of the marketed oral oseltamivir suspension dosed according to the HD or CAPD schedule, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (>/=) 18 years of age
* ESRD defined as no residual renal function or a creatinine clearance (CrCl) less than (<) 10 milliliters per minute (mL/min)
* Well established HD or CAPD therapy over a period of 3 months with stable CrCl < 10 mL/min
* Body mass index (BMI) 18 to 34 kilograms per meter-squared (kg/m^2)
* Use of contraception among women of childbearing potential

Exclusion Criteria:

* Clinical significant comorbid disease or terminal illness
* Known human immunodeficiency virus (HIV) or hepatitis B or C
* History of drug or alcohol abuse within the prior year
* Donation or loss of >/= 400 milliliters (mL) of blood in the 3 months prior to Screening
* Participation in a clinical study with an investigational drug in the 3 months prior to study drug
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-10; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- Oseltamivir With HD: Participants on hemodialysis (HD) received 9 doses of 30-milligram (mg) oseltamivir oral suspension, given 1 hour after completion of alternating HD sessions. All HD participants were planned to receive 19 routine HD sessions (three per week) during the 6.5-week study period.
- Oseltamivir With CAPD: Participants on continuous ambulatory peritoneal dialysis (CAPD) received 6 doses of 30-mg oseltamivir oral suspension, given once weekly after dialysis exchange. All CAPD participants underwent routine CAPD sessions (four exchanges per 24 hours) during the 6-week study period.
Period: Overall Study
Arm/Group | Oseltamivir With HD | Oseltamivir With CAPD
Started | 12 (None were prematurely withdrawn; 1 switched to CAPD mid-study and was excluded from second analysis.) | 12
First Dose Assessment Period | 12 | 12
Second Dose Assessment Period | 11 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled: All participants enrolled into the study regardless of treatment received.
Groups:
- Oseltamivir With HD: Participants on HD received 9 doses of 30-mg oseltamivir oral suspension, given 1 hour after completion of alternating HD sessions. All HD participants were planned to receive 19 routine HD sessions (three per week) during the 6.5-week study period.
- Oseltamivir With CAPD: Participants on CAPD received 6 doses of 30-mg oseltamivir oral suspension, given once weekly after dialysis exchange. All CAPD participants underwent routine CAPD sessions (four exchanges per 24 hours) during the 6-week study period.
- Total: Total of all reporting groups
Arm/Group | Oseltamivir With HD | Oseltamivir With CAPD | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.00 (13.23) | 54.42 (14.30) | 51.21 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 11 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Oseltamivir in HD Participants During Days 1 to 5
Description: Plasma samples were obtained up to 90 hours post-dose during the first dose analysis (Days 1 to 5), and the maximum observed concentration was recorded. The Cmax was averaged among all participants and expressed in nanograms per milliliter (ng/mL).
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from Day 1 (D1) dose
Population: Pharmacokinetic (PK) Analysis Population (First Dose Subpopulation): All participants who completed treatment and provided evaluable data during the first dose assessment period.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng/mL | 20.2 (12.3)

2. Primary Outcome: Cmax of Oseltamivir in HD Participants During Days 38 to 43
Description: Plasma samples were obtained up to 90 hours post-dose during the second dose analysis (Days 38 to 43), and the maximum observed concentration was recorded. The Cmax was averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from Day 38 (D38) dose
Population: PK Analysis Population (Second Dose Subpopulation): All participants who completed treatment and provided evaluable data during the second dose assessment period.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 11
ng/mL | 22.6 (9.69)

3. Primary Outcome: Cmax of Metabolite Oseltamivir Carboxylate in HD Participants During Days 1 to 5
Description: Plasma samples were obtained up to 90 hours post-dose during the first dose analysis (Days 1 to 5), and the maximum observed concentration was recorded. The Cmax was averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng/mL | 943 (393)

4. Primary Outcome: Cmax of Metabolite Oseltamivir Carboxylate in HD Participants During Days 38 to 43
Description: as for outcome 2
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D38 dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 11
ng/mL | 1120 (320)

5. Primary Outcome: Area Under the Concentration-Time Curve (AUC) of Oseltamivir in HD Participants During Days 1 to 5
Description: Plasma samples were obtained up to 90 hours post-dose during the first dose analysis (Days 1 to 5), and the AUC was determined from 0 to 12 hours (AUC12) and up to the last measurable concentration (AUClast). Values were averaged among all participants and expressed in nanograms by hours per milliliter (ng*h/mL).
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng*h/mL
  AUC12 | 63.9 (24.6)
  AUClast | 62.1 (26.8)

6. Primary Outcome: AUC of Oseltamivir in HD Participants During Days 38 to 43
Description: Plasma samples were obtained up to 90 hours post-dose during the second dose analysis (Days 38 to 43), and the AUC12 and AUClast were determined. Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D38 dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 11
ng*h/mL
  AUC12 | 68.5 (19.5)
  AUClast | 65.6 (20.1)

7. Primary Outcome: AUC of Metabolite Oseltamivir Carboxylate in HD Participants During Days 1 to 5
Description: Plasma samples were obtained up to 90 hours post-dose during the first dose analysis (Days 1 to 5), and the AUC was determined from 0 to 42 hours (AUC42) and up to the last measurable concentration (AUClast). Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng*h/mL
  AUC42 | 31600 (14100)
  AUClast | 44400 (19000)

8. Primary Outcome: AUC of Metabolite Oseltamivir Carboxylate in HD Participants During Days 38 to 43
Description: Plasma samples were obtained up to 90 hours post-dose during the second dose analysis (Days 38 to 43), and the AUC42 and AUClast were determined. Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D38 dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 11
ng*h/mL
  AUC42 | 38200 (11500)
  AUClast | 60400 (16700)

9. Primary Outcome: Cmax of Oseltamivir in CAPD Participants During Days 1 to 6
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6), and the maximum observed concentration was recorded. The Cmax was averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng/mL | 32.0 (20.4)

10. Primary Outcome: Cmax of Oseltamivir in CAPD Participants During Days 36 to 43
Description: Plasma samples were obtained up to 168 hours post-dose during the second dose analysis (Days 36 to 43), and the maximum observed concentration was recorded. The Cmax was averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168 hours from Day 36 (D36) dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng/mL | 27.7 (15.9)

11. Primary Outcome: Cmax of Metabolite Oseltamivir Carboxylate in CAPD Participants During Days 1 to 6
Description: as for outcome 9
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng/mL | 885 (244)

12. Primary Outcome: Cmax of Metabolite Oseltamivir Carboxylate in CAPD Participants During Days 36 to 43
Description: as for outcome 10
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168 hours from D36 dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng/mL | 849 (200)

13. Primary Outcome: AUC of Oseltamivir in CAPD Participants During Days 1 to 6
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6), and the AUC12 and AUClast were determined. Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng*h/mL
  AUC12 | 85.6 (40.7)
  AUClast | 78.5 (41.8)

14. Primary Outcome: AUC of Oseltamivir in CAPD Participants During Days 36 to 43
Description: Plasma samples were obtained up to 168 hours post-dose during the second dose analysis (Days 36 to 43), and the AUC12 and AUClast were determined. Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168 hours from D36 dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng*h/mL
  AUC12 | 72.4 (28.3)
  AUClast | 67.7 (27.7)

15. Primary Outcome: AUC of Metabolite Oseltamivir Carboxylate in CAPD Participants During Days 1 to 6
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6), and the AUC was determined from 0 to 48 hours (AUC48) and up to the last measurable concentration (AUClast). Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng*h/mL
  AUC48 | 33400 (9700)
  AUClast | 56800 (18300)

16. Primary Outcome: AUC of Metabolite Oseltamivir Carboxylate in CAPD Participants During Days 36 to 43
Description: Plasma samples were obtained up to 168 hours post-dose during the second dose analysis (Days 36 to 43), and the AUC48 and AUClast were determined. Values were averaged among all participants and expressed in ng*h/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168 hours from D36 dose
Population: PK Analysis Population (Second Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng*h/mL
  AUC48 | 32400 (8210)
  AUClast | 60800 (18800)

17. Secondary Outcome: Plasma Concentration of Oseltamivir by Timepoint in HD Participants
Description: Plasma samples were obtained up to 90 hours post-dose during the first dose analysis (Days 1 to 5) and up to 114 hours post-dose during the second dose analysis (Days 38 to 43). The concentration at each collection time was recorded and averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49 hours from D1 and D38 dose AND at 90 hours from D1 dose AND at 114 hours from D38 dose
Population: PK Analysis Population; number (n) equals (=) number of participants included at specified timepoints in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng/mL
  0 hours from D1 dose (n=12) | 0 (0)
  1 hour from D1 dose (n=12) | 18.0 (14.2)
  2 hours from D1 dose (n=12) | 12.5 (6.58)
  4 hours from D1 dose (n=12) | 6.06 (2.37)
  8 hours from D1 dose (n=12) | 1.93 (1.64)
  12 hours from D1 dose (n=12) | 0.513 (0.783)
  20 hours from D1 dose (n=12) | 0.104 (0.361)
  32 hours from D1 dose (n=12) | 0.0 (0.0)
  42 hours from D1 dose (n=12) | 0.0 (0.0)
  48 hours from D1 dose (n=12) | 0.0 (0.0)
  49 hours from D1 dose (n=12) | 0.0 (0.0)
  90 hours from D1 dose (n=12) | 0.0 (0.0)
  0 hours from D38 dose (n=11) | 0.413 (0.938)
  1 hour from D38 dose (n=11) | 21.5 (9.96)
  2 hours from D38 dose (n=11) | 15.4 (5.98)
  4 hours from D38 dose (n=11) | 6.07 (2.80)
  8 hours from D38 dose (n=11) | 1.30 (0.801)
  12 hours from D38 dose (n=11) | 0.193 (0.429)
  20 hours from D38 dose (n=11) | 0.0 (0.0)
  32 hours from D38 dose (n=11) | 0.0 (0.0)
  42 hours from D38 dose (n=11) | 0.0 (0.0)
  48 hours from D38 dose (n=11) | 0.0 (0.0)
  49 hours from D38 dose (n=11) | 0.0 (0.0)
  114 hours from D38 dose (n=11) | 0.0 (0.0)

18. Secondary Outcome: Plasma Concentration of Metabolite Oseltamivir Carboxylate by Timepoint in HD Participants
Description: as for outcome 17
Time Frame: as for outcome 17
Population: PK Analysis Population; n = number of participants included at specified timepoints in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng/mL
  0 hours from D1 dose (n=12) | 0.908 (3.15)
  1 hour from D1 dose (n=12) | 25.7 (24.5)
  2 hours from D1 dose (n=12) | 107 (83.7)
  4 hours from D1 dose (n=12) | 276 (181)
  8 hours from D1 dose (n=12) | 589 (321)
  12 hours from D1 dose (n=12) | 772 (363)
  20 hours from D1 dose (n=12) | 908 (383)
  32 hours from D1 dose (n=12) | 926 (399)
  42 hours from D1 dose (n=12) | 877 (393)
  48 hours from D1 dose (n=12) | 212 (78.6)
  49 hours from D1 dose (n=12) | 233 (88.2)
  90 hours from D1 dose (n=12) | 240 (123)
  0 hours from D38 dose (n=11) | 59.0 (32.1)
  1 hour from D38 dose (n=11) | 95.0 (32.8)
  2 hours from D38 dose (n=11) | 200 (58.7)
  4 hours from D38 dose (n=11) | 413 (137)
  8 hours from D38 dose (n=11) | 745 (239)
  12 hours from D38 dose (n=11) | 933 (295)
  20 hours from D38 dose (n=11) | 1090 (327)
  32 hours from D38 dose (n=11) | 1080 (328)
  42 hours from D38 dose (n=11) | 1050 (340)
  48 hours from D38 dose (n=11) | 263 (61.4)
  49 hours from D38 dose (n=11) | 279 (66.4)
  114 hours from D38 dose (n=11) | 283 (112)

19. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Oseltamivir in HD Participants
Description: Plasma samples were obtained up to 90 hours post-dose during the first (Days 1 to 5) and second (Days 38 to 43) dose analyses, and the observed time of maximum concentration was recorded. The Tmax following each dose was averaged among all participants and expressed in hours.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D1 and D38 dose
Population: PK Analysis Population; n = number of participants included in the specific dose analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
hours
  Days 1 to 5 (n=12) | 1.75 (1.14)
  Days 38 to 43 (n=11) | 1.18 (0.40)

20. Secondary Outcome: Tmax of Metabolite Oseltamivir Carboxylate in HD Participants
Description: as for outcome 19
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from D1 and D38 dose
Population: PK Analysis Population; n = number of participants included in the specific dose analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
hours
  Days 1 to 5 (n=12) | 29.7 (8.0)
  Days 38 to 43 (n=11) | 29.2 (9.61)

21. Secondary Outcome: Oral Plasma Clearance (CL/F) of Oseltamivir in HD Participants
Description: Plasma samples up to 12 hours post-dose during the first (Days 1 to 5) and second (Days 38 to 43) dose analyses were used to calculate apparent clearance adjusted for oral bioavailability. The CL/F with each dose was averaged among all participants and expressed in liters per hour (L/h).
Time Frame: Blood samples 0, 1, 2, 4, 8, 12 hours from D1 and D38 dose
Population: PK Analysis Population; n = number of participants included in the specific dose analysis.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
L/h
  Days 1 to 5 (n=12) | 677 (727)
  Days 38 to 43 (n=11) | 474 (141)

22. Secondary Outcome: CL/F of Metabolite Oseltamivir Carboxylate in HD Participants
Description: Plasma samples up to 42 hours post-dose during the first (Days 1 to 5) and second (Days 38 to 43) dose analyses were used to calculate apparent clearance adjusted for oral bioavailability. The CL/F with each dose was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42 hours from D1 and D38 dose
Population: PK Analysis Population; n = number of participants included in the specific dose analysis.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
L/h
  Days 1 to 5 (n=12) | 1.20 (1.05)
  Days 38 to 43 (n=11) | 0.779 (0.239)

23. Secondary Outcome: Renal Clearance (CLr) of Oseltamivir in HD Participants
Description: Plasma and urine samples up to 12 hours post-dose during the first dose analysis (Days 1 to 5) were used to calculate CLr, computed as [amount of drug excreted divided by the AUC12]. The CLr was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12 hours from D1 dose; urine samples 0 to 12 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
L/h | 0.0521 (0.133)

24. Secondary Outcome: CLr of Metabolite Oseltamivir Carboxylate in HD Participants
Description: Plasma and urine samples up to 42 hours post-dose during the first dose analysis (Days 1 to 5) were used to calculate CLr, computed as [amount of metabolite excreted divided by the AUC42]. The CLr was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42 hours from D1 dose; urine samples 0 to 42 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
L/h | 0.0203 (0.0568)

25. Secondary Outcome: Dialysis Clearance (CLd) of Metabolite Oseltamivir Carboxylate in HD Participants
Description: Plasma samples up to 90 hours post-dose during the first (Days 1 to 5) and second (Days 38 to 43) dose analyses, in addition to dialyzer samples obtained on Days 3 and 40, were used to calculate CLd, computed as [amount of metabolite recovered in dialysate divided by the AUC over the dialysis interval]. The CLd with each dose was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 20, 32, 42, 48, 49, 90 hours from from D1 and D38 dose; dialyzer samples 1, 2, 4, 5 hours from start of dialysis on Days 3 and 40
Population: PK Analysis Population; n = number of participants included in the specific dose analysis.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
L/h
  Days 1 to 5 (n=12) | 7.42 (0.447)
  Days 38 to 43 (n=11) | 8.43 (3.02)

26. Secondary Outcome: Percentage of Oseltamivir Dose Excreted as Unchanged Drug in HD Participants
Description: Urine samples up to 42 hours post-dose during the first dose analysis (Days 1 to 5) were used to calculate drug excretion, computed as [amount of drug excreted divided by the oral oseltamivir dose] multiplied by 100. The value was averaged among all participants and expressed as a percent of the oseltamivir dose administered.
Time Frame: Urine samples 0 to 42 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: percentage of oseltamivir dose
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
percentage of oseltamivir dose | 0.00982 (0.0221)

27. Secondary Outcome: Percentage of Oseltamivir Dose Excreted as Metabolite Oseltamivir Carboxylate in HD Participants
Description: Urine samples up to 42 hours post-dose during the first dose analysis (Days 1 to 5) were used to calculate metabolite excretion, computed as [amount of metabolite excreted divided by the oral oseltamivir dose] multiplied by 100. The value was averaged among all participants and expressed as a percent of the oseltamivir dose administered.
Time Frame: Urine samples 0 to 42 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: percentage of osteltamivir dose
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
percentage of osteltamivir dose | 1.86 (4.66)

28. Secondary Outcome: Plasma Concentration of Metabolite Oseltamivir Carboxylate in Arterial and Venous Blood by Timepoint in HD Participants
Description: Dialyzer samples were obtained up to 5 hours from the start of dialysis on Days 3 and 40 (corresponding to HD sessions 2 and 18). Arterial concentrations were estimated using the inflow to the dialyzer, and venous concentrations were estimated using the outflow from the dialyzer. The concentration at each collection time was recorded and averaged among all participants and expressed in ng/mL.
Time Frame: Dialyzer samples 1, 2, 4, 5 hours from start of dialysis on Days 3 and 40
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With HD
Number analyzed (Participants) | 12
ng/mL
  Arterial: 1 hour (Day 3) | 570 (229)
  Arterial: 2 hours (Day 3) | 412 (157)
  Arterial: 4 hours (Day 3) | 227 (82.2)
  Arterial: 5 hours (Day 3) | 171 (61.8)
  Venous: 1 hour (Day 3) | 284 (121)
  Venous: 2 hours (Day 3) | 202 (74.4)
  Venous: 4 hours (Day 3) | 127 (69.1)
  Venous: 5 hours (Day 3) | 84.3 (29.6)
  Arterial: 1 hour (Day 40) | 666 (179)
  Arterial: 2 hours (Day 40) | 496 (125)
  Arterial: 4 hours (Day 40) | 281 (58.8)
  Arterial: 5 hours (Day 40) | 218 (45.6)
  Venous: 1 hour (Day 40) | 317 (103)
  Venous: 2 hours (Day 40) | 229 (69.6)
  Venous: 4 hours (Day 40) | 128 (37.3)
  Venous: 5 hours (Day 40) | 95.4 (27.7)

29. Secondary Outcome: Plasma Concentration of Oseltamivir by Timepoint in CAPD Participants
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6) and up to 168 hours post-dose during the second dose analysis (Days 36 to 43). The concentration at each collection time was recorded and averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 and D36 dose AND at 168 hours from D36 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng/mL
  0 hours from D1 dose | 0.0 (0.0)
  1 hour from D1 dose | 27.8 (21.9)
  2 hours from D1 dose | 22.6 (12.6)
  4 hours from D1 dose | 6.98 (2.70)
  8 hours from D1 dose | 0.630 (0.833)
  12 hours from D1 dose | 0.100 (0.346)
  24 hours from D1 dose | 0.0 (0.0)
  48 hours from D1 dose | 0.0 (0.0)
  72 hours from D1 dose | 0.0 (0.0)
  120 hours from D1 dose | 0.0 (0.0)
  0 hours from D36 dose | 0.0 (0.0)
  1 hour from D36 dose | 24.8 (16.8)
  2 hours from D36 dose | 18.0 (8.88)
  4 hours from D36 dose | 5.78 (2.09)
  8 hours from D36 dose | 0.754 (0.705)
  12 hours from D36 dose | 0.103 (0.358)
  24 hours from D36 dose | 0.0 (0.0)
  48 hours from D36 dose | 0.0 (0.0)
  72 hours from D36 dose | 0.0 (0.0)
  120 hours from D36 dose | 0.0 (0.0)
  168 hours from D36 dose | 0.0 (0.0)

30. Secondary Outcome: Plasma Concentration of Metabolite Oseltamivir Carboxylate by Timepoint in CAPD Participants
Description: Plasma samples were obtained up to 120 post-dose during the first dose analysis (Days 1 to 6) and up to 168 hours post-dose during the second dose analysis (Days 36 to 43). The concentration at each collection time was recorded and averaged among all participants and expressed in ng/mL.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 and D36 dose AND at 168 hours from D36 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
ng/mL
  0 hours from D1 dose | 0.0 (0.0)
  1 hour from D1 dose | 20.3 (19.9)
  2 hours from D1 dose | 121 (72.7)
  4 hours from D1 dose | 381 (171)
  8 hours from D1 dose | 691 (217)
  12 hours from D1 dose | 812 (251)
  24 hours from D1 dose | 879 (245)
  48 hours from D1 dose | 580 (193)
  72 hours from D1 dose | 360 (148)
  120 hours from D1 dose | 147 (80.9)
  0 hours from D36 dose | 69.2 (40.1)
  1 hour from D36 dose | 97.0 (52.3)
  2 hours from D36 dose | 184 (84.7)
  4 hours from D36 dose | 403 (149)
  8 hours from D36 dose | 663 (179)
  12 hours from D36 dose | 802 (200)
  24 hours from D36 dose | 831 (201)
  48 hours from D36 dose | 563 (172)
  72 hours from D36 dose | 362 (138)
  120 hours from D36 dose | 149 (71.6)
  168 hours from D36 dose | 63.0 (38.1)

31. Secondary Outcome: Tmax of Oseltamivir in CAPD Participants
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6) and up to 168 hours post-dose during the second dose analysis (Days 36 to 43), and the observed time of maximum concentration was recorded. The Tmax following each dose was averaged among all participants and expressed in hours.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 and D36 dose AND at 168 hours from D36 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
hours
  Days 1 to 6 | 1.50 (0.52)
  Days 36 to 43 | 1.28 (0.0470)

32. Secondary Outcome: Tmax of Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: as for outcome 31
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 and D36 dose AND at 168 hours from D36 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
hours
  Days 1 to 6 | 20.0 (5.91)
  Days 36 to 43 | 19.0 (6.18)

33. Secondary Outcome: Elimination Rate Constant of Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6) and up to 168 hours post-dose during the second dose analysis (Days 36 to 43). Urine and dialysate samples were also obtained up to 48 hours post-dose during the first dose analysis. The elimination rate constant was calculated as [natural log (ln)(2) divided by the half-life] and expressed as inverse hours (1/h).
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 and D36 dose AND at 168 hours from D36 dose; urine samples 0 to 48 hours from D1 dose; dialysate samples 0 to 48 hours from D1 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
1/h
  Days 1 to 6 | 0.0211 (0.00578)
  Days 36 to 43 | 0.0200 (0.00488)

34. Secondary Outcome: Terminal Elimination Half-Life of Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Plasma samples were obtained up to 120 hours post-dose during the first dose analysis (Days 1 to 6) and up to 168 hours post-dose during the second dose analysis (Days 36 to 43). Urine and dialysate samples were also obtained up to 48 hours post-dose during the first dose analysis. The time required for the concentration to decrease by one-half was recorded and averaged among all participants and expressed in hours.
Time Frame: as for outcome 33
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
hours
  Days 1 to 6 | 34.8 (8.39)
  Days 36 to 43 | 36.3 (7.53)

35. Secondary Outcome: CL/F of Oseltamivir in CAPD Participants
Description: Plasma samples up to 12 hours post-dose during the first (Days 1 to 6) and second (Days 36 to 43) dose analyses were used to calculate apparent clearance adjusted for oral bioavailability. The CL/F with each dose was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12 hours from D1 and D36 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
L/h
  Days 1 to 6 | 424 (183)
  Days 36 to 43 | 485 (215)

36. Secondary Outcome: CL/F of Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Plasma samples up to 48 hours post-dose during the first (Days 1 to 6) and second (Days 36 to 43) dose analyses were used to calculate apparent clearance adjusted for oral bioavailability. The CL/F with each dose was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48 hours from D1 and D36 dose
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
L/h
  Days 1 to 6 | 0.882 (0.250)
  Days 36 to 43 | 0.898 (0.246)

37. Secondary Outcome: CLr of Oseltamivir in CAPD Participants
Description: Plasma and urine samples up to 12 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate CLr, computed as [amount of drug excreted divided by the AUC12]. The CLr was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12 hours from D1 dose; urine samples 0 to 12 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
L/h | 0.146 (0.250)

38. Secondary Outcome: CLr of Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Plasma and urine samples up to 48 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate CLr, computed as [amount of metabolite excreted divided by the AUC48]. The CLr was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48 hours from D1 dose; urine samples 0 to 48 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
L/h | 0.0665 (0.114)

39. Secondary Outcome: CLd of Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Plasma samples up to 120 hours and dialysate samples up to 48 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate CLd, computed as [amount of metabolite recovered in dialysate divided by the AUC over the dialysis interval]. The CLd was averaged among all participants and expressed in L/h.
Time Frame: Blood samples 0, 1, 2, 4, 8, 12, 24, 48, 72, 120 hours from D1 dose; dialysate samples 0 to 48 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
L/h | 0.425 (0.0456)

40. Secondary Outcome: Percentage of Oseltamivir Dose Renally Excreted as Unchanged Drug in CAPD Participants
Description: Urine samples up to 48 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate renal excretion, computed as [amount of drug in urine divided by the oral oseltamivir dose] multiplied by 100. The value was averaged among all participants and expressed as a percent of the oseltamivir dose administered.
Time Frame: Urine samples 0 to 48 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: percentage of oseltamivir dose
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
percentage of oseltamivir dose | 0.0290 (0.0490)

41. Secondary Outcome: Percentage of Oseltamivir Dose Renally Excreted as Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Urine samples up to 48 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate renal excretion, computed as [amount of metabolite in urine divided by the oral oseltamivir dose] multiplied by 100. The value was averaged among all participants and expressed as a percent of the oseltamivir dose administered.
Time Frame: Urine samples 0 to 48 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: percentage of oseltamivir dose
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
percentage of oseltamivir dose | 6.44 (10.8)

42. Secondary Outcome: Percentage of Oseltamivir Dose Eliminated by Dialysis as Unchanged Drug in CAPD Participants
Description: Dialysate samples up to 48 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate dialysis elimination, computed as [amount of drug in dialysate divided by the oral oseltamivir dose] multiplied by 100. The value was averaged among all participants and expressed as a percent of the oseltamivir dose administered.
Time Frame: Dialysate samples 0 to 48 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: percentage of oseltamivir dose
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
percentage of oseltamivir dose | 0.00367 (0.0127)

43. Secondary Outcome: Percentage of Oseltamivir Dose Eliminated by Dialysis as Metabolite Oseltamivir Carboxylate in CAPD Participants
Description: Dialysate samples up to 48 hours post-dose during the first dose analysis (Days 1 to 6) were used to calculate dialysis elimination, computed as [amount of metabolite in dialysate divided by the oral oseltamivir dose] multiplied by 100. The value was averaged among all participants and expressed as a percent of the oseltamivir dose administered.
Time Frame: Dialysate samples 0 to 48 hours from D1 dose
Population: PK Analysis Population (First Dose Subpopulation).
Measure: Mean (Standard Deviation); unit: percentage of oseltamivir dose
Arm/Group | Oseltamivir With CAPD
Number analyzed (Participants) | 12
percentage of oseltamivir dose | 32.6 (8.77)

ADVERSE EVENTS:
Time Frame: From Day 1 to 43 and up to 14 days after last PK assessment (up to approximately 57 days total)
Description: Safety Population
Arm/Group | Oseltamivir With HD | Oseltamivir With CAPD
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/12
Other Adverse Events (participants affected / at risk) | 8/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir With HD (N=12) | Oseltamivir With CAPD (N=12)
Angina unstable (Cardiac disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericarditis not otherwise specified (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir With HD (N=12) | Oseltamivir With CAPD (N=12)
Vomiting not otherwise specified (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 3
Diarrhoea not otherwise specified (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Dizziness (excluding vertigo) (General disorders) | 2 | 0
Malaise (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Haemorrhage not otherwise specified (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Pain in jaw (General disorders) | 0 | 1
Headache not otherwise specified (Nervous system disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Appetite decreased (Metabolism and nutrition disorders) | 0 | 1
Calcification metastatic (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder not otherwise specified (Skin and subcutaneous tissue disorders) | 0 | 1
Tongue oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat not otherwise specified (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood culture positive (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Urinary tract infection not otherwise specified (Infections and infestations) | 0 | 1
Vaginitis (Infections and infestations) | 0 | 1
Vaginosis bacterial not otherwise specified (Infections and infestations) | 0 | 1
Anaemia not otherwise specified (Blood and lymphatic system disorders) | 0 | 1
Anaemia not otherwise specified, aggravated (Blood and lymphatic system disorders) | 0 | 1
Hepatic function abnormal not otherwise specified (Hepatobiliary disorders) | 0 | 1
Skin injury not otherwise specified (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Depression not otherwise specified (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.